CLINICAL TRIAL: NCT01578473
Title: An Open-Label, Nine-Month Randomized Controlled Study of Testosterone (Testopel) Pellets Plus Vitamin D and E Versus Vitamin D and E Alone for the Treatment of Peyronie's Disease
Brief Title: Testosterone Pellets Plus Vitamin D and E Versus Vitamin D and E Alone for the Treatment of Peyronie's Disease
Acronym: PD+
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Men's Health Boston (Other)
Responsible Party: Principal Investigator, Dr. Abraham Morgentaler, Associate Clinical Professor of Urology Harvard Medical School, Men's Health Boston
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: PD Plus Study; SAIRB #201107293 (Other: Schulman Associates Institutional Review Board, Inc.)
Record Dates: First submitted 2012-04-12; First posted 2012-04-17 (Estimated); Last update posted 2018-03-29 (Actual); Status verified 2018-03

CONDITIONS: Peyronie's Disease
Keywords: low testosterone; penile curvature
MeSH Terms: conditions — Penile Induration | interventions — Ergocalciferols; Vitamin E; Testosterone

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Vitamin D and E (Active Comparator): Oral Vitamin D and E alone in men with penile curvature due to PD.
  Interventions: Drug: Vitamin D2; Drug: Vitamin E
- Testosterone Pellets and Vitamin D and E (Active Comparator): Testosterone in combination with oral Vitamin D an E supplementation in men with penile curvature due to PD.
  Interventions: Drug: Testosterone Pellets

INTERVENTIONS:
Drug: Vitamin D2 — oral softgel 2000 IU once daily 9 months
  Other Names: 21st Century Dietary Supplement
  Arms: Vitamin D and E
Drug: Vitamin E — oral softgels 400 IU and 200 IU 1 softgel of 400 IU daily
  1 softgel of 200 IU daily 9 months
  Other Names: GERI-CARE
  Arms: Vitamin D and E
Drug: Testosterone Pellets — subcutaneous implantation pellets 75 mg based on testosterone levels from resulting bloodwork 9 months
  Other Names: Testopel 75 mg testosterone pellets
  Arms: Testosterone Pellets and Vitamin D and E

SUMMARY:
Two recent studies have identified low levels of serum testosterone in association with Peyronie's Disease (PD), with a significant correlation noted between severity of testosterone deficiency and severity of curvature. The study hypothesis is to determine whether treatment with testosterone may help men with PD and penile curvature.

ELIGIBILITY:
Inclusion Criteria:

* acquired penile curvature of > 30 degrees and < 90 degrees associated with palpable penile plaque on physical examination
* onset of curvature within 18 months prior to signing consent form
* serum TT < 500 ng/dl at the screening visit

Exclusion Criteria:

* prior history of treatment for PD that includes intra-lesional injections, topical creams, or surgery
* prior treatment with oral therapy at least 2 weeks prior to signing consent form (e.g. Potaba, Vitamin E, colchicines) will be acceptable for inclusion
* prior history of treatment for testosterone deficiency
* presence of dense calcified plaque by US or plain radiograph
* taking the medication Coumadin
* hypersensitivity to testosterone, stearic acid, or polyvinyl pyrolidone (the constituents of Testopel)
* unable to achieve adequate erection with penile injection to access degree of curvature
* undergone definitive treatment for prostate cancer, bladder cancer, or other pelvic malignancies including surgery, external beam radiation therapy, brachytherapy, cryotherapy.
* prior history of prostate cancer, hematologic disorders, chronic liver disease including cirrhosis and hepatitis C, disorders affecting the immune system, including infection with human immunodeficiency virus, or psychiatric disorders including major depression, schizophrenia, bipolar disease
* history of cerebrovascular accident, history of deep venous thrombosis within the past 5 years or history of untreated or severe sleep apnea
* PSA > 4.0 ng/dL at the screening visit, unless prostate cancer has been excluded to the investigator's satisfaction
* clinically significant abnormal lab results that would put the subject at increased risk or compromise the integrity of the study data, in the opinion of the investigator
* received any other investigational drug within 30 days

Ages: 18 Years to 70 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 75 (Actual)
Dates: Start 2013-05-23 (Actual); Primary Completion 2013-07-07 (Actual); Study Completion 2017-11-13 (Actual)

PRIMARY OUTCOMES:
penile curvature | 9 months
  The primary outcome to be assessed will be the change in penile curvature from baseline.

SECONDARY OUTCOMES:
sexual function | 9 months
  Secondary outcomes will incluce overall satisfaction with sexual function (patient satisfaction with treatment, quality of erections and quality of life).

CONTACTS AND LOCATIONS:
Overall Officials: Abraham Morgentaler, MD, Principal Investigator — Men's Health Boston
Locations (1):
- Men's Health Boston, Chestnut Hill, Massachusetts, United States